CLINICAL TRIAL: NCT01364454
Title: Effect of Eligible Patients Paper-based Reminder for General Practitioners on Colorectal Cancer Screening Participation
Brief Title: General Practitioners (GP) Involvement in Colorectal Cancer (CRC) Screening
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Paris 12 Val de Marne University (Other)
Responsible Party: Principal Investigator, Julien Le Breton, MD, MPH, Paris 12 Val de Marne University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DUERMG
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Screening; Faecal Occult Blood test; General Practitioners Involvement; Patient's Participation; Reminder
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eligible patients' paper-based reminder (Experimental)
  Interventions: Other: Eligible patients' paper-based reminder
- Control group (No Intervention)

INTERVENTIONS:
Other: Eligible patients' paper-based reminder — Providing to the general practitioners every four months a list of their patients who are eligible for colorectal cancer screening but did not proceed yet and were not excluded for medical reason
  Arms: Eligible patients' paper-based reminder

SUMMARY:
Screening for ColoRectal Cancer (CRC) is widely recommended because of compelling evidence that it reduces mortality from CRC and that it's cost-effective. In France, there is a national CRC screening programme inviting people aged 50-74 years by mail to consult their General Practitioner (GP) for a free on charge Faecal Occult Blood test deliverance every two years. Participation is a key factor for the screening programs success. High levels of screening uptake and the continued participation to regular screening must be achieved and maintained in the targeted population if the enormous potential of CRC screening is to be realised. Screening rates of various international programs vary widely (20-52%) and the participation is insufficient in the most settings. Therefore, a better understanding of facilitating and hindering factors of patient participation can guide interventions to improve CRC screening rates. They include patients and physicians' factors. One issue is about GPs practice. GP involvement has been shown to improve the participation in the CRC screening. This study aims to assess the effectiveness of an intervention targeting GPs to increase patient participation in the CRC screening. Volunteer GPs will be randomly assigned to either the intervention group or to usual care (control group) and they will be followed one year. The intervention consists in providing every four months to the experimental group a list of their patients who are eligible but did not proceed yet to the screening. In both groups, patient participation in the screening will be measured at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. General Practitioner (GP)

   * exercising in the Val de Marne (French department of the suburb of Paris)
   * volunteered to participate at the study
2. Patient

   * living in the Val de Marne (French department of the suburb of Paris)
   * having declared a 'preferred GP' exercising in the Val de Marne to the main statutory health insurance scheme ("régime général")
   * being eligible for colorectal cancer screening (aged 50 to 74 years, not excluded and having not proceed yet to the screening)
   * having consulted his 'preferred GP', whatever the reason, during the study period

Exclusion Criteria:

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8140 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Patient's participation to colorectal cancer screening program | 1 year
  Patient's status with colorectal cancer screening program to 15th june 2011 with two modalities
  1. Update: completion of Faecal Occult Blood test or exclusion for medical reason within the duration of the study (The medical exclusions of the program are a personal or family history of Colorectal cancer, Crohn's disease, hemorrhagic rectocolitis, or hereditary nonpolyposis colorectal cancer, a colonoscopy undergone in the 5 previous years or a Fecal Occult Blood test undergone in the 2 previous years)
  2. Not update

CONTACTS AND LOCATIONS:
Overall Officials: Julien Le Breton, MD, MPH, Principal Investigator — DUERMG
Locations (1):
- Département Universitaire d'Enseignement et de Recherche en Médecine Générale, Créteil, France